CLINICAL TRIAL: NCT07150247
Title: A Phase II Single-Arm Study of Iparomlimab and Tuvonralimab Combined With Bevacizumab and FOLFIRI in BRAF V600E-Mutant Metastatic Colorectal Cancer
Brief Title: Safety and Efficacy of IB-FOLFIRI in BRAF V600E-Mutant Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Deshen Wang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IB-FOLFIRI
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: BRAF V600 Colorectal Cancer
Keywords: Objective response rate; Circulating tumor DNA; Phase II clinical trial; BRAF V600E colorectal cancer
MeSH Terms: interventions — Bevacizumab; Fluorouracil; Irinotecan; Pharmaceutical Preparations

STUDY DESIGN:
Intervention Model Description: Prospecitve Single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Iparomlimab and Tuvonralimab+ Bevacizumab + FOLFIRI (Experimental): Given every two weeks
  Interventions: Drug: Iparomlimab and Tuvonralimab; Drug: Bevacizumab; Drug: 5-Fluorouracil; Drug: Irinotecan (drug)

INTERVENTIONS:
Drug: Iparomlimab and Tuvonralimab — 3mg/kg，ivdrip
  Other Names: QL1706
Drug: Bevacizumab — 5mg/kg，ivdrip
  Other Names: Avastin
Drug: 5-Fluorouracil — 400mg/m2 iv followed by 2.4g/m2 civ 48h
  Other Names: 5-FU
Drug: Irinotecan (drug) — 180mg/m2
  Other Names: CPT-11

SUMMARY:
The goal of this clinical trial is to learn if Iparomlimab and Tuvonralimab combined with bevacizumab and FOLFIRI (IB-FOLFIRI) is safe and effective in treating adults with BRAF V600E-mutant metastatic colorectal cancer (mCRC). The main questions it aims to answer are:

Does IB-FOLFIRI improve clinical outcomes compared with historical outcomes in this population?

What is the safety profile of IB-FOLFIRI in patients with BRAF V600E-mutant mCRC?

Participants will:

Receive Iparomlimab and Tuvonralimab, bevacizumab, and FOLFIRI every two weeks

Have blood samples and/or tumor tissue collected for biomarker analysis (e.g., ctDNA sequencing)

Undergo regular imaging and clinical evaluations to assess treatment response and safety

DETAILED DESCRIPTION:
This is a single-arm, phase II clinical trial designed to evaluate the safety and efficacy of Iparomlimab and Tuvonralimab plus bevacizumab combined with FOLFIRI (IB-FOLFIRI) in patients with BRAF V600E-mutant metastatic colorectal cancer (mCRC). Patients with this genetic subtype have limited treatment options and a poor prognosis, underscoring the urgent need for more effective therapeutic strategies.

This study will generate prospective clinical data on the efficacy and safety of the IB-FOLFIRI regimen in a genetically defined subgroup of colorectal cancer. Furthermore, exploratory biomarker analyses may provide new insights into resistance mechanisms, potentially guiding future precision-medicine strategies for BRAF V600E-mutant mCRC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years
* Histologically confirmed metastatic colorectal adenocarcinoma
* BRAF V600E mutation confirmed by tissue pathology or ctDNA testing (PCR or NGS)
* Disease progression after at least one line of treatment: FOLFOX/XELOX (oxaliplatin-based doublet) ± bevacizumab or FOLFOXIRI (irinotecan-based triplet) ± bevacizumab. Note: Irinotecan must not have failed during prior treatment, and disease must not have progressed within three months of stopping treatment
* Patients who have received first-line treatment with cetuximab combined with a BRAF inhibitor (e.g., encorafenib, dabrafenib, vemurafenib) are allowed
* At least one measurable lesion according to RECIST v1.1 criteria
* Adequate hematologic unction: Platelets > 90 × 10⁹/L; Hemoglobin > 100 g/L; White blood cells > 3 × 10⁹/L; Neutrophils > 1.5 × 10⁹/L; Adequate liver function; Total bilirubin ≤ 1.5 × ULN; AST and ALT ≤ 2.5 × ULN (≤ 5 × ULN if liver metastases present); Alkaline phosphatase ≤ 2.5 × ULN; No ascites; Coagulation: PT ≤ 1.5 × ULN, INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN, Albumin ≥ 30 g/L
* Adequate renal function: CrCl ≥ 50 mL/min or serum creatinine ≤ 1.5 × ULN
* Liver function Child-Pugh class A
* ECOG performance status 0-1
* Expected survival > 3 months
* Signed written informed consent
* Willing and able to comply with follow-up until death, study completion, or study termination
* For women of childbearing potential: Negative serum pregnancy test within 14 days prior to treatment; Willing to use medically accepted contraception during the study and for 3 months after the last dose
* For male participants with partners of childbearing potential: Must have undergone surgical sterilization, or use effective contraception during the study and for 3 months after the last dose

Exclusion Criteria:

* KRAS or NRAS mutation
* MSI-H/dMMR patients
* Prior treatment with PD-1, PD-L1, or CTLA-4 inhibitors
* Known contraindications to irinotecan at the planned dose
* Use of systemic immunosuppressive drugs within 1 week prior to treatment
* Active autoimmune disease requiring treatment, or history of such disease within the past 2 years
* Known primary immunodeficiency
* History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation
* Retinal vein occlusion or risk factors for retinal vein occlusion (e.g., uncontrolled glaucoma or high intraocular pressure)
* History of acute or chronic pancreatitis
* Chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory, immunosuppressive therapy, or surgery) within 12 months prior to enrollment
* Gastrointestinal disorders that may significantly affect oral drug absorption (e.g., severe GI ulcers, uncontrolled vomiting, malabsorption syndrome, short bowel syndrome)
* Neuromuscular diseases associated with elevated CK (e.g., inflammatory myopathy, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
* Residual ≥Grade 2 toxicity from prior anti-tumor therapy (excluding ≥Grade 2 alopecia or neuropathy)
* History of HIV infection
* History of Gilbert's syndrome
* Interstitial pneumonia or extensive symptomatic interstitial pulmonary fibrosis
* Severe uncontrolled systemic comorbidities
* Severe cardiovascular disease, including:
* Stroke within 6 months prior to enrollment
* Myocardial infarction within 6 months prior to enrollment
* Hypertension not controlled with appropriate medications
* Unstable angina
* Congestive heart failure (NYHA class 2-4)
* Cardiac arrhythmias requiring treatment
* Current or prior central nervous system disease, including: Primary brain tumor; Epilepsy not controlled by standard treatment; Any brain metastases or history of stroke
* Other uncontrolled comorbidities, including active bleeding, uncontrolled infection or non-malignant medical conditions that could be worsened by study therapy, or uncontrolled psychiatric/social conditions
* History of other malignancies within the past 5 years (except for curatively treated basal cell carcinoma, cervical carcinoma in situ, or thyroid cancer)
* Allergy to any study drug
* Pregnant or breastfeeding women
* Women of childbearing potential (last menstrual period <2 years) or men who refuse to use effective non-hormonal contraception (IUD, barrier method plus spermicide, or sterilization)
* Inability or unwillingness to comply with study protocol
* Any other disease, metastatic lesion-related functional impairment, or suspicious findings on physical examination that may indicate contraindication to study drug use or place the patient at high risk of treatment-related complications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Assessed after every 4 cycles (each cycle is 2 weeks) from treatment initiation until radiographic disease progression, treatment discontinuation, or completion of the 3-year follow-up, whichever occurs first
  The percentage of patients in a study group who have a partial or complete response to treatment according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Progression Free Survival | Assessed throughout the study duration (3 years)
  The proportion of patients who remain alive and whose disease does not progress after starting treatment
Overall survival | Assessed throughout the study duration (5 years)
  Time from treatment initiation to death from any cause or censored due to loss to follow up
Adverse events | Assessed throughout the study duration (3 years)
  Assessment of adverse events and their severity according to NCI CTCAE version 5.0 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
Data and materials used in this study can be made available following study completion upon reasonable request to the corresponding author, subject to ethical and legal considerations and applicable data-sharing agreements.